CLINICAL TRIAL: NCT01927341
Title: A Phase Ib/II, Open-label, Multi-center, Dose Escalation Study of MEK162 in Combination With Panitumumab in Adult Patients With Mutant RAS or Wild-type RAS Metastatic Colorectal Cancer
Brief Title: Phase Ib/II Study of Efficacy and Safety of MEK162 and Panitumumab, in Adult mCRC Patients With Mutant or Wild-type RAS Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CMEK162X2116; C4211008 (Other: Alias Study Number); 2013-001986-18 (EudraCT Number)
Record Dates: First submitted 2013-08-02; First posted 2013-08-22 (Estimated); Results first posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-01

CONDITIONS: Metastatic Colorectal Cancer
Keywords: MEK162,; panitumumab,; mutant RAS,; wild-type RAS,; metastatic colorectal cancer,; adult mCRC patient
MeSH Terms: conditions — Colorectal Neoplasms | interventions — binimetinib; Panitumumab

ARMS (5):
- Phase Ib: Dose escalation (Experimental): Phase Ib: Dose escalation.
  Interventions: Drug: MEK162; Drug: Panitumumab
- Phase II: Patients with mutant RAS mCRC (Experimental): Patients with mutant RAS mCRC who have not been pretreated with an EGFR inhibitor (EGFRi), including EGFR tyrosine kinase inhibitor therapy and/or anti-EGFR monoclonal antibody therapy.
  Interventions: Drug: MEK162; Drug: Panitumumab
- Phase II: Patients with acquired mutant RAS mCRC (Experimental): Patients with acquired mutant RAS mCRC who have been pretreated with anti-EGFR monoclonal antibody therapy, but have not been pre-treated with EGFR tyrosine kinase inhibitor therapy.
  Interventions: Drug: MEK162; Drug: Panitumumab
- Phase II: Patients with WT RAS mCRC (pretreated) (Experimental): Patients with WT RAS mCRC who have been pretreated with an EGFRi, including EGFR tyrosine kinase inhibitor therapy and/or anti-EGFR monoclonal antibody therapy.
  Interventions: Drug: MEK162; Drug: Panitumumab
- Phase II: Patients with WT RAS mCRC (not pretreated) (Experimental): Patients with WT RAS mCRC who have not been pretreated with an EGFRi, including EGFR tyrosine kinase inhibitor therapy and/or anti-EGFR monoclonal antibody therapy.
  Interventions: Drug: MEK162; Drug: Panitumumab

INTERVENTIONS:
Drug: MEK162 — Tablet for oral use, 45 mg (three 15 mg tablets), BID
Drug: Panitumumab — Intravenous infusion, 20mg/ml concentrate solution for infusion, Q2W (Days 1 and 15 of every cycle)

SUMMARY:
The primary purpose of the phase Ib is to estimate the MTD/RPD2 and of the phase II is to assess the anti-tumor activity of MEK162 in combination with panitumumab.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Metastatic colorectal cancer
* Progression on or following standard therapy, or no standard therapy (phase Ib). Progression on or following at least 2-prior fluoropyrimidine-containing chemotherapy regimens (phase II)
* Written documentation of mutant or wild-type RAS
* Life expectancy ≥ 3 months
* ECOG performance status ≤ 2

Exclusion Criteria:

Phase II arms 1 and 4 only: previous treatment with cetuximab, panitumumab, and/or other EGFR inhibitors

* Previous treatment with MEK-inhibitors
* History of severe infusion reactions to monoclonal antibodies.
* Symptomatic or untreated leptomeningeal disease
* Symptomatic brain metastasis
* Current evidence of retinal disease; history of CSR, RVO or ophthalmopathy as assessed by ophthalmologic examination at baseline that would be considered a risk factor for CSR/RVO and history of keratitis.
* Acute or chronic pancreatitis
* Clinically significant cardiac disease
* Not adequate hematologic, renal and hepatic function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2013-11-19 (Actual); Primary Completion 2016-01-25 (Actual); Study Completion 2016-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- United States (2):
  - University of California at Los Angeles Dept of Onc, Los Angeles, California
  - Memorial Sloan Kettering Cancer Center Oncology Dept, New York, New York
- Pfizer Investigative Site, Leuven, Belgium
- Pfizer Investigative Site, Toronto, Ontario, Canada
- Pfizer Investigative Site, Toulouse, France
- Pfizer Investigative Site, Milan, MI, Italy
- Pfizer Investigative Site, Amsterdam, Netherlands
- Pfizer Investigative Site, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Van Cutsem E, Yaeger R, Delord JP, Tabernero J, Siu LL, Ducreux M, Siena S, Elez E, Kasper S, Zander T, Steeghs N, Murphy D, Edwards M, Wainberg ZA. Phase Ib/II Study of the Efficacy and Safety of Binimetinib (MEK162) Plus Panitumumab for Mutant or Wild-Type RAS Metastatic Colorectal Cancer. Oncologist. 2023 Dec 11;28(12):e1209-e1218. doi: 10.1093/oncolo/oyad210. PMID 37597246

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study had Phase 1b followed by Phase 2. Phase 1b was to evaluate the maximum tolerated dose (MTD)/recommended Phase 2 dose (RPD2) in participants with mutant or wild type (WT) rat sarcoma viral oncogene homologue (RAS) metastatic colorectal cancer (mCRC) who had progressed on or following standard therapy or for whom no standard therapy existed. Phase 2 assessed anti-tumor activity in participants enrolled based on the previous anti-EGFR monoclonal antibody therapy and RAS mutational status.
Pre-assignment Details: The study used binimetinib 45 mg twice a day (BID) and panitumumab 6 mg/kg intravenous infusion once every second week without planned dose escalation.
Groups:
- Phase 1b: Binimetinib (MEK162) + Panitumumab: Participants received binimetinib 45 milligram (mg) orally twice daily with panitumumab 6 milligram per kilogram (mg/kg) intravenous (IV) infusion once every second week on Days 1 and 15 of every cycle (1 cycle = 28 days) until progression of disease, unacceptable toxicity develops, or withdrawal of informed consent, whichever occurred first. Maximum treatment exposure was approximately of 40 weeks.
- Phase 2:Mutant RAS Epidermal Growth Factor Receptor Inhibitor(EGFRi)-Naive:Binimetinib + Panitumumab: Participants with mutant RAS mCRC who had not been pretreated with an EGFRi, including EGFR tyrosine kinase inhibitor therapy and/or anti-EGFR monoclonal antibody therapy, received binimetinib 45 mg orally twice daily with panitumumab 6 mg/kg IV infusion once every second week on Days 1 and 15 of every cycle (1 cycle = 28 days) until progression of disease, unacceptable toxicity develops, or withdrawal of informed consent, whichever occurred first. Maximum treatment exposure was approximately of 15.4 weeks.
- Phase 2: Mutant RAS Anti-EGFRi: Binimetinib + Panitumumab: Participants with acquired mutant RAS mCRC who had been pretreated with anti-EGFR monoclonal antibody therapy, but had not been pre-treated with EGFR tyrosine kinase inhibitor therapy, received binimetinib 45 mg orally twice daily with panitumumab 6 mg/kg IV infusion once every second week on Days 1 and 15 of every cycle (1 cycle = 28 days) until progression of disease, unacceptable toxicity develops, or withdrawal of informed consent, whichever occurred first. Maximum treatment exposure was approximately of 33.7 weeks.
- Phase 2: WT RAS Anti-EGFRi: Binimetinib + Panitumumab: Participants with WT RAS mCRC who had been pretreated with an anti-EGFRi monoclonal antibody therapy but had not been pretreated with EGFR tyrosine kinase inhibitor therapy, received binimetinib 45 mg orally twice daily with panitumumab 6 mg/kg IV infusion once every second week on Days 1 and 15 of every cycle (1 cycle = 28 days) until progression of disease, unacceptable toxicity develops, or withdrawal of informed consent, whichever occurred first. Maximum treatment exposure was approximately of 32.1 weeks.
- Phase 2: WT RAS EGFRi-Naive: Binimetinib + Panitumumab: Participants with WT RAS mCRC who had not been pretreated with an EGFRi, including EGFR tyrosine kinase inhibitor therapy and/or anti-EGFR monoclonal antibody therapy, received binimetinib 45 mg orally twice daily with panitumumab 6 mg/kg IV infusion once every second week on Days 1 and 15 of every cycle (1 cycle = 28 days) until progression of disease, unacceptable toxicity develops, or withdrawal of informed consent, whichever occurred first. Maximum treatment exposure was approximately of 48.0 weeks.
Period: Phase 1b
Arm/Group | Phase 1b: Binimetinib (MEK162) + Panitumumab | Phase 2:Mutant RAS Epidermal Growth Factor Receptor Inhibitor(EGFRi)-Naive:Binimetinib + Panitumumab | Phase 2: Mutant RAS Anti-EGFRi: Binimetinib + Panitumumab | Phase 2: WT RAS Anti-EGFRi: Binimetinib + Panitumumab | Phase 2: WT RAS EGFRi-Naive: Binimetinib + Panitumumab
Started | 10 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 10 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Death | 2 | 0 | 0 | 0 | 0
Not completed — Follow-up completed | 7 | 0 | 0 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1b: Binimetinib (MEK162) + Panitumumab | Phase 2:Mutant RAS Epidermal Growth Factor Receptor Inhibitor(EGFRi)-Naive:Binimetinib + Panitumumab | Phase 2: Mutant RAS Anti-EGFRi: Binimetinib + Panitumumab | Phase 2: WT RAS Anti-EGFRi: Binimetinib + Panitumumab | Phase 2: WT RAS EGFRi-Naive: Binimetinib + Panitumumab
Started | 0 | 15 (Participants of phase 2 enrolled after enrollment of participants of phase 1b.) | 5 (Participants of phase 2 enrolled after enrollment of participants of phase 1b.) | 15 (Participants of phase 2 enrolled after enrollment of participants of phase 1b.) | 8 (Participants of phase 2 enrolled after enrollment of participants of phase 1b.)
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 15 | 5 | 15 | 8
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Participant withdrew consent | 0 | 2 | 1 | 2 | 3
Not completed — Death | 0 | 4 | 0 | 3 | 2
Not completed — New cancer therapy | 0 | 1 | 0 | 4 | 1
Not completed — Disease progression | 0 | 1 | 1 | 1 | 0
Not completed — Follow-up completed | 0 | 6 | 3 | 5 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who received at least 1 full or partial dose of study drug.
Groups:
- Phase 1b: Binimetinib + Panitumumab: Participants received binimetinib 45 mg orally twice daily with panitumumab 6 mg/kg IV infusion once every second week on Days 1 and 15 of every cycle (1 cycle = 28 days) until progression of disease, unacceptable toxicity develops, or withdrawal of informed consent, whichever occurred first. Maximum treatment exposure was approximately of 40 weeks.
- Phase 2: Mutant RAS EGFRi-Naive: Binimetinib + Panitumumab: Participants with mutant RAS mCRC who had not been pretreated with an EGFRi, including EGFR tyrosine kinase inhibitor therapy and/or anti-EGFR monoclonal antibody therapy, received binimetinib 45 mg orally twice daily with panitumumab 6 mg/kg IV infusion once every second week on Days 1 and 15 of every cycle (1 cycle = 28 days) until progression of disease, unacceptable toxicity develops, or withdrawal of informed consent, whichever occurred first. Maximum treatment exposure was approximately of 15.4 weeks.
- Total: Total of all reporting groups
Arm/Group | Phase 1b: Binimetinib + Panitumumab | Phase 2: Mutant RAS EGFRi-Naive: Binimetinib + Panitumumab | Phase 2: Mutant RAS Anti-EGFRi: Binimetinib + Panitumumab | Phase 2: WT RAS Anti-EGFRi: Binimetinib + Panitumumab | Phase 2: WT RAS EGFRi-Naive: Binimetinib + Panitumumab | Total
Number analyzed (Participants) | 10 | 15 | 5 | 15 | 8 | 53
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.1 (10.6) | 54.3 (11.2) | 60.2 (12.0) | 59.8 (14.0) | 54.1 (10.7) | 56.4 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 4 | 9 | 5 | 31
  Male | 6 | 6 | 1 | 6 | 3 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLT): Phase 1b
Description: DLT was defined as an adverse event or clinically significant abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurred within the first 28 days of treatment (Cycle 1) with binimetinib and panitumumab and met any of the specified criteria.
Time Frame: Within the first 28 days of treatment with binimetinib and panitumumab (Cycle 1)
Population: Dose determining set included all phase 1b participants who received at least 1 dose of binimetinib or panitumumab and had at least 1 valid post baseline safety assessment, and those who had either experienced a DLT at any time during Cycle 1 or had met the following minimum treatment and safety evaluation requirements without experiencing a DLT during Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Binimetinib + Panitumumab
Number analyzed (Participants) | 10
Participants | 0

2. Primary Outcome: Overall Response Rate (ORR) as Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 Based on Local Radiology Assessment: Phase 2
Description: ORR: percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR) as assessed per RECIST version 1.1. BOR: the best response recorded from the start of the treatment until CR or PR. CR: disappearance of all non-nodal target lesions and of all non-target lesions. In addition, any pathological lymph nodes assigned as target lesions/ non-target lesions must have a reduction in short axis to <10 mm. PR: at least a 30 percent (%) decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: From the start of the treatment until CR or PR (approximately up to 11 months)
Population: Full analysis set included all participants who received at least 1 full or partial dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Phase 2: Mutant RAS EGFRi-Naive: Binimetinib + Panitumumab | Phase 2: Mutant RAS Anti-EGFRi: Binimetinib + Panitumumab | Phase 2: WT RAS Anti-EGFRi: Binimetinib + Panitumumab | Phase 2: WT RAS EGFRi-Naive: Binimetinib + Panitumumab
Number analyzed (Participants) | 15 | 5 | 15 | 8
Percentage of participants | 0 [0 to 0] | 0 [0 to 0] | 6.7 [0.2 to 31.9] | 0 [0 to 0]

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAE)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline (Day 1) up to 28 days after last dose of study drug (approximately up to 12 months)
Population: Safety analysis set included all participants who received at least 1 full or partial dose of study drug and had at least 1 valid post-baseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Binimetinib + Panitumumab | Phase 2: Mutant RAS EGFRi-Naive: Binimetinib + Panitumumab | Phase 2: Mutant RAS Anti-EGFRi: Binimetinib + Panitumumab | Phase 2: WT RAS Anti-EGFRi: Binimetinib + Panitumumab | Phase 2: WT RAS EGFRi-Naive: Binimetinib + Panitumumab
Number analyzed (Participants) | 10 | 15 | 5 | 15 | 8
Participants
  TEAEs | 10 | 15 | 5 | 15 | 8
  SAEs | 3 | 6 | 2 | 9 | 5

4. Secondary Outcome: Number of Participants With Vital Sign Abnormalities
Description: Vital sign abnormalities criteria included: 1) Systolic blood pressure (SBP) in millimeters of mercury (mmHg): greater than or equal to (>=)180 mmHg or less than equal to (<=) 90 mmHg with increase or decrease from baseline of >=20 mmHg with high and low post baseline values; 2) Diastolic blood pressure (DBP) (mmHg): >=105 mmHg or <=50 mmHg with increase or decrease from baseline of >=15 mmHg with high and low post baseline values; 3) Pulse rate in beats per minutes (bpm): >=120 bpm or <=50 bpm with increase or decrease from baseline of >=15 bpm with high and low post baseline values; 4) Weight in kilogram: >=10% increase or decrease from baseline with high and low post baseline values; 5) Oral body temperature in degree Celsius (C) : >=39 degree C or <=35 degree C with high and low post baseline values. Categories, with at least 1 participant having vital sign abnormality in any of the reporting arms, were reported in this outcome measure.
Time Frame: Baseline (Day 1) up to 28 days after last dose of study drug (approximately up to 12 months)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Binimetinib + Panitumumab | Phase 2: Mutant RAS EGFRi-Naive: Binimetinib + Panitumumab | Phase 2: Mutant RAS Anti-EGFRi: Binimetinib + Panitumumab | Phase 2: WT RAS Anti-EGFRi: Binimetinib + Panitumumab | Phase 2: WT RAS EGFRi-Naive: Binimetinib + Panitumumab
Number analyzed (Participants) | 10 | 15 | 5 | 15 | 8
Participants
  SBP :>=180 mmHg or <=90 mmHg with increase or decrease from baseline of >=20 mmHg: low only | 0 | 1 | 1 | 2 | 0
  DBP: >=105 mmHg or <=50 mmHg with increase or decrease from baseline of >=15 mmHg: high only | 0 | 1 | 0 | 0 | 0
  Pulse: >=120 bpm or <=50 bpm with increase or decrease from baseline of >=15 bpm: high only | 0 | 3 | 1 | 2 | 1
  Pulse:>=120 bpm or <=50 bpm with increase or decrease from baseline of >=15 bpm: low only | 0 | 0 | 0 | 1 | 0
  Weight: >=10 % increase or decrease from baseline: high only | 0 | 1 | 0 | 1 | 0
  Weight: >=10 % increase or decrease from baseline: low only | 1 | 0 | 0 | 1 | 0
  Oral body temperature: >=39 °C or <=35 °C: high only | 1 | 0 | 0 | 0 | 0
  Oral body temperature: >=39 °C or <=35 °C: low only | 0 | 0 | 1 | 0 | 1

5. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: ECG abnormalities criteria included: 1) QTc interval adjusted according to Bazett formula (QTcB) in millisecond (msec): greater than (>) 450, >480, >500, increase from baseline >30, increase from baseline >60; 2) QTc interval adjusted according to Fridericia formula (QTcF) (msec): >450, >480, >500, increase from baseline >30, increase from baseline >60; 3) Heart rate (bpm): RR decrease >25% and to a VR (interval between QRS wave and T wave on ECG) >100; RR (interval between 2 successive R waves on ECG) increase >25% and to a VR <50; 4) Pulse rate (msec): increase >25% and to a value >200; 5) QT (msec): >450, >480, >500, increase from baseline >30, increase from baseline >60; 6) QRS (msec): increase >25% and to a value >110. Categories, with at least 1 participant having ECG abnormality in any of the reporting arms, were reported in this outcome measure.
Time Frame: Baseline (Day 1) up to 28 days after last dose of study drug (approximately up to 12 months)
Population: Safety analysis set included all participants who received at least 1 full or partial dose of study drug and had at least 1 valid post-baseline safety assessment. Here, "number analyzed" signifies participants evaluable at specific rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Binimetinib + Panitumumab | Phase 2: Mutant RAS EGFRi-Naive: Binimetinib + Panitumumab | Phase 2: Mutant RAS Anti-EGFRi: Binimetinib + Panitumumab | Phase 2: WT RAS Anti-EGFRi: Binimetinib + Panitumumab | Phase 2: WT RAS EGFRi-Naive: Binimetinib + Panitumumab
Number analyzed (Participants) | 10 | 15 | 5 | 15 | 8
Participants
  QTcB: >450 msec: number analyzed (Participants) | 8 | 13 | 5 | 12 | 5
  QTcB: >450 msec | 3 | 2 | 1 | 5 | 1
  QTcB: >480 msec: number analyzed (Participants) | 10 | 15 | 5 | 14 | 6
  QTcB: >480 msec | 1 | 1 | 0 | 2 | 0
  QTcB: >500 msec: number analyzed (Participants) | 10 | 15 | 5 | 14 | 6
  QTcB: >500 msec | 0 | 1 | 0 | 0 | 0
  QTcB: Increase from baseline >30 msec: number analyzed (Participants) | 10 | 15 | 5 | 14 | 6
  QTcB: Increase from baseline >30 msec | 3 | 5 | 1 | 1 | 2
  QTcF: >450 msec: number analyzed (Participants) | 10 | 15 | 5 | 13 | 6
  QTcF: >450 msec | 1 | 1 | 0 | 1 | 2
  QTcF: Increase from baseline >30 msec: number analyzed (Participants) | 10 | 15 | 5 | 14 | 6
  QTcF: Increase from baseline >30 msec | 3 | 2 | 1 | 1 | 1
  Heart rate: RR decrease >25% and to a VR >100 bpm: number analyzed (Participants) | 10 | 15 | 5 | 14 | 6
  Heart rate: RR decrease >25% and to a VR >100 bpm | 1 | 1 | 0 | 1 | 0
  Heart rate: RR increase >25% and to a VR <50 bpm: number analyzed (Participants) | 10 | 15 | 5 | 14 | 6
  Heart rate: RR increase >25% and to a VR <50 bpm | 0 | 1 | 0 | 0 | 0
  QT: >450 msec: number analyzed (Participants) | 10 | 15 | 5 | 14 | 5
  QT: >450 msec | 0 | 1 | 0 | 1 | 1
  QT: >480 msec: number analyzed (Participants) | 10 | 15 | 5 | 14 | 6
  QT: >480 msec | 0 | 1 | 0 | 0 | 0
  QT: increase from baseline >30 msec: number analyzed (Participants) | 10 | 15 | 5 | 14 | 6
  QT: increase from baseline >30 msec | 6 | 3 | 1 | 5 | 4
  QT: increase from baseline >60 msec: number analyzed (Participants) | 10 | 15 | 5 | 14 | 6
  QT: increase from baseline >60 msec | 0 | 2 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Following parameters were analyzed for laboratory examination: hematology (hematocrit, erythrocytes); biochemistry (direct bilirubin, blood urea nitrogen, calcium, creatine kinase, triiodothyronine, thyroxine and thyrotropin). Clinical significance of laboratory abnormalities were judged by investigator.
Time Frame: Baseline (Day 1) up to 28 days after last dose of study drug (approximately up to 12 months)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Binimetinib + Panitumumab | Phase 2: Mutant RAS EGFRi-Naive: Binimetinib + Panitumumab | Phase 2: Mutant RAS Anti-EGFRi: Binimetinib + Panitumumab | Phase 2: WT RAS Anti-EGFRi: Binimetinib + Panitumumab | Phase 2: WT RAS EGFRi-Naive: Binimetinib + Panitumumab
Number analyzed (Participants) | 10 | 15 | 5 | 15 | 8
Participants | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Overall Response Rate (ORR) as Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 Based on Local Radiology Assessment: Phase 1b
Description: as for outcome 2
Time Frame: From the start of the treatment until disease progression (approximately up to 11 months)
Population: Full analysis set included all participants who received at least 1 full or partial dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Phase 1b: Binimetinib + Panitumumab
Number analyzed (Participants) | 10
Percentage of participants | 0 [0 to 0]

8. Secondary Outcome: Progression-free Survival (PFS) as Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 Based on Local Radiology Assessment
Description: PFS: time from date of randomization to date of first documented PD or death due to any cause, whichever occurred first. RECIST 1.1, PD:>=20% increase in sum of diameter of all measured target lesions (TLs), taking as reference smallest sum of diameter of all TLs recorded at or after baseline, sum must also be absolute increase of >=5 mm^2. Unequivocal progression of existing non-TLs. Appearance of new lesions. With no event at time of analysis cut-off or at start of any new anti-neoplastic therapy, PFS was censored at date of last adequate tumor assessment of complete response (CR), partial response (PR) or stable disease (SD). CR:disappearance of all non-nodal TLs/non TLs, any pathological lymph nodes as TLs/non TLs must have reduction in short axis to <10 mm. PR:>=30% decrease in sum of diameter of all TLs, referring baseline sum of diameters. SD:neither sufficient shrinkage to qualify for PR or CR nor increase in lesions qualified for PD. Kaplan-Meier method used for PFS analysis.
Time Frame: From the date of randomization to the date of the first documented PD or death (approximately up to 11 months)
Population: Full analysis set included all participants who received at least 1 full or partial dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1b: Binimetinib + Panitumumab | Phase 2: Mutant RAS EGFRi-Naive: Binimetinib + Panitumumab | Phase 2: Mutant RAS Anti-EGFRi: Binimetinib + Panitumumab | Phase 2: WT RAS Anti-EGFRi: Binimetinib + Panitumumab | Phase 2: WT RAS EGFRi-Naive: Binimetinib + Panitumumab
Number analyzed (Participants) | 10 | 15 | 5 | 15 | 8
Months | 3.4 [1.4 to 5.2] | 1.7 [1.5 to 3.4] | 1.8 [1.6 to 8.2] | 2.4 [1.6 to 3.5] | 2.1 [1.0 to 10.8]

9. Secondary Outcome: Duration of Response (DOR) as Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 Based on Local Radiology Assessment
Description: DOR: time from first documented occurrence of response (PR or CR) until date of first documented PD or death due to underlying cancer. RECIST 1.1. CR: disappearance of all non-nodal target lesions and of all non-target lesions. In addition, any pathological lymph nodes assigned as target lesions/ non-target lesions must have a reduction in short axis to <10 mm. PR: at least a 30% decrease in sum of diameter of all target lesions, taking as reference baseline sum of diameters. PD: at least a 20% increase in sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, sum must also demonstrate an absolute increase of at least 5 mm^2. Unequivocal progression of existing non-target lesions. Appearance of new lesions. Participants with no PD and were still alive, were censored at last adequate tumor assessment. Kaplan-Meier method was used for DOR analysis.
Time Frame: From the first documented occurrence of response (PR or CR) until the date of the first documented PD or death due to the underlying cancer (approximately up to 11 months)
Population: Full analysis set included all participants who received at least 1 full or partial dose of study drug. The outcome was to be analyzed only in confirmed responders, none of the reporting arms had confirmed responders except Phase 2: WT RAS Anti-EGFRi: Binimetinib + Panitumumab.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1b: Binimetinib + Panitumumab | Phase 2: Mutant RAS EGFRi-Naive: Binimetinib + Panitumumab | Phase 2: Mutant RAS Anti-EGFRi: Binimetinib + Panitumumab | Phase 2: WT RAS Anti-EGFRi: Binimetinib + Panitumumab | Phase 2: WT RAS EGFRi-Naive: Binimetinib + Panitumumab
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
Months |  |  |  | 5.3 [NA to NA] — Lower and upper limit of confidence interval was not estimable due to low number of participants with an event. |

10. Secondary Outcome: Disease Control Rate (DCR) as Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 Based on Local Radiology Assessment
Description: DCR was defined as the percentage of participants with a confirmed BOR of CR, PR, or stable disease (SD). RECIST 1.1, BOR was defined as the best response recorded from the start of the treatment until CR, PR or SD. CR: disappearance of all non-nodal target lesions and of all non-target lesions. In addition, any pathological lymph nodes assigned as target lesions/ non-target lesions must have a reduction in short axis to <10 mm. PR: at least a 30 percent (%) decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. PD: at least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm^2. Unequivocal progression of existing non-target lesions. Appearance of new lesions.
Time Frame: From the start of the treatment until disease progression (approximately up to 11 months)
Population: Full analysis set included all participants who received at least 1 full or partial dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1b: Binimetinib + Panitumumab | Phase 2: Mutant RAS EGFRi-Naive: Binimetinib + Panitumumab | Phase 2: Mutant RAS Anti-EGFRi: Binimetinib + Panitumumab | Phase 2: WT RAS Anti-EGFRi: Binimetinib + Panitumumab | Phase 2: WT RAS EGFRi-Naive: Binimetinib + Panitumumab
Number analyzed (Participants) | 10 | 15 | 5 | 15 | 8
Percentage of participants | 70.0 [34.8 to 93.3] | 13.3 [1.7 to 40.5] | 40.0 [5.3 to 85.3] | 40.0 [16.3 to 67.7] | 37.5 [8.5 to 75.5]

11. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the start of treatment to the date of death due to any cause. If a participant was not known to have died, survival was censored at the date of last known date patient alive. Kaplan-Meier method was used for OS analysis.
Time Frame: From the start of treatment to the date of death due to any cause (approximately up to 11 months)
Population: Full analysis set included all participants who received at least 1 full or partial dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1b: Binimetinib + Panitumumab | Phase 2: Mutant RAS EGFRi-Naive: Binimetinib + Panitumumab | Phase 2: Mutant RAS Anti-EGFRi: Binimetinib + Panitumumab | Phase 2: WT RAS Anti-EGFRi: Binimetinib + Panitumumab | Phase 2: WT RAS EGFRi-Naive: Binimetinib + Panitumumab
Number analyzed (Participants) | 10 | 15 | 5 | 15 | 8
Months | NA [1.9 to NA] — Median and lower limit of confidence interval was not estimable due to low number of participants with an event. | 3.5 [2.1 to 8.0] | 5.5 [3.9 to 9.6] | 5.8 [3.1 to 8.0] | 11.2 [2.1 to 13.3]

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last dose of study drug (approximately up to 12 months)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety analysis set included all the participants who received at least 1 dose of study drug and had at least 1 valid post-baseline safety assessment.
Arm/Group | Phase 1b: Binimetinib + Panitumumab | Phase 2: Mutant RAS EGFRi-Naive: Binimetinib + Panitumumab | Phase 2: Mutant RAS Anti-EGFRi: Binimetinib + Panitumumab | Phase 2: WT RAS Anti-EGFRi: Binimetinib + Panitumumab | Phase 2: WT RAS EGFRi-Naive: Binimetinib + Panitumumab
Serious Adverse Events (participants affected / at risk) | 3/10 | 6/15 | 2/5 | 9/15 | 5/8
Other Adverse Events (participants affected / at risk) | 10/10 | 15/15 | 5/5 | 15/15 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Binimetinib + Panitumumab (N=10) | Phase 2: Mutant RAS EGFRi-Naive: Binimetinib + Panitumumab (N=15) | Phase 2: Mutant RAS Anti-EGFRi: Binimetinib + Panitumumab (N=5) | Phase 2: WT RAS Anti-EGFRi: Binimetinib + Panitumumab (N=15) | Phase 2: WT RAS EGFRi-Naive: Binimetinib + Panitumumab (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1
General Physical Health Deterioration (General disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Septic Shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Skin Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 0 | 0 | 1 | 0
Platelet Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Troponin T Increased (Investigations) | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypovolaemic Shock (Vascular disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Binimetinib + Panitumumab (N=10) | Phase 2: Mutant RAS EGFRi-Naive: Binimetinib + Panitumumab (N=15) | Phase 2: Mutant RAS Anti-EGFRi: Binimetinib + Panitumumab (N=5) | Phase 2: WT RAS Anti-EGFRi: Binimetinib + Panitumumab (N=15) | Phase 2: WT RAS EGFRi-Naive: Binimetinib + Panitumumab (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 4 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 3 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 2 | 2 | 1 | 2 | 0
Chorioretinopathy (Eye disorders) | 2 | 0 | 0 | 4 | 0
Retinal Detachment (Eye disorders) | 1 | 0 | 2 | 1 | 1
Retinopathy (Eye disorders) | 2 | 1 | 0 | 1 | 1
Periorbital Oedema (Eye disorders) | 2 | 0 | 0 | 1 | 0
Vitreous Floaters (Eye disorders) | 1 | 1 | 0 | 0 | 1
Dry Eye (Eye disorders) | 1 | 0 | 0 | 1 | 0
Eye Swelling (Eye disorders) | 1 | 0 | 0 | 1 | 0
Eye Discharge (Eye disorders) | 1 | 0 | 0 | 0 | 0
Iritis (Eye disorders) | 1 | 0 | 0 | 0 | 0
Visual Impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 9 | 5 | 13 | 4
Vomiting (Gastrointestinal disorders) | 4 | 8 | 4 | 9 | 3
Nausea (Gastrointestinal disorders) | 5 | 8 | 4 | 5 | 5
Abdominal Pain (Gastrointestinal disorders) | 1 | 3 | 4 | 4 | 2
Stomatitis (Gastrointestinal disorders) | 3 | 1 | 0 | 6 | 3
Constipation (Gastrointestinal disorders) | 2 | 4 | 1 | 5 | 0
Dry Mouth (Gastrointestinal disorders) | 1 | 5 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 1 | 2 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 2
Oral Pain (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Gastrointestinal Inflammation (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 9 | 5 | 1 | 5 | 5
Chills (General disorders) | 3 | 3 | 1 | 1 | 2
Oedema Peripheral (General disorders) | 2 | 4 | 2 | 1 | 1
Pyrexia (General disorders) | 2 | 4 | 1 | 3 | 0
Asthenia (General disorders) | 0 | 2 | 0 | 5 | 1
Feeling Cold (General disorders) | 3 | 0 | 0 | 0 | 0
Face Oedema (General disorders) | 1 | 0 | 0 | 0 | 0
Facial Pain (General disorders) | 1 | 0 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 0 | 0 | 0
Peripheral Swelling (General disorders) | 1 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 3 | 0 | 1 | 3 | 1
Folliculitis (Infections and infestations) | 0 | 2 | 0 | 3 | 0
Conjunctivitis (Infections and infestations) | 1 | 1 | 0 | 2 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 2 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 2 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Rash Pustular (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Skin Infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Septic Shock (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Stoma Site Pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 5 | 3 | 2 | 6 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 3 | 1 | 4 | 0
Ejection Fraction Decreased (Investigations) | 1 | 2 | 2 | 1 | 1
Blood Creatinine Increased (Investigations) | 0 | 1 | 0 | 5 | 0
Lipase Increased (Investigations) | 1 | 1 | 2 | 1 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 2 | 1 | 2 | 0
Blood Bilirubin Increased (Investigations) | 0 | 2 | 1 | 1 | 0
Weight Decreased (Investigations) | 3 | 0 | 1 | 0 | 0
Amylase Increased (Investigations) | 1 | 0 | 1 | 0 | 1
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 2 | 0 | 1 | 0
Intraocular Pressure Increased (Investigations) | 1 | 0 | 0 | 1 | 0
Troponin Increased (Investigations) | 1 | 0 | 0 | 1 | 0
Haemoglobin Decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 2 | 0 | 4 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 5 | 1 | 1 | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 5 | 1 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 1 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 3 | 0 | 1 | 1 | 1
Neuropathy Peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Retinal Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0
Genital Haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 8 | 5 | 1 | 4 | 5
Rash (Skin and subcutaneous tissue disorders) | 2 | 7 | 2 | 9 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 6 | 1 | 1 | 4 | 5
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 5 | 0 | 1 | 2 | 4
Skin Fissures (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 3 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Nail Disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Swelling Face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Trichorrhexis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 3 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 1 | 0 | 0
Vasculitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Fungal Skin Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study used binimetinib 45 mg BID and panitumumab 6 mg/kg intravenous infusion once every second week, there was no planned dose escalation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.